CLINICAL TRIAL: NCT02976779
Title: A Phase I, Double Blind, Randomized, Placebo Controlled, Maximal Dose Study to Determine the Safety, Tolerability of Topical Cream Containing MGC (Medical Grade Cannabis) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: One World Cannabis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OWC-PSO-01
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-01

CONDITIONS: Safety Study for Future Treatment of Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OWC MGC cream (Experimental): Cannabis based topical cream 3% CBD and 3% THC. The cream was designed to treat Psoriasis . The cream will be applied twice daily.
  Interventions: Drug: OWC MGC cream
- OWC Control Cream (Placebo Comparator): Carrier cream. CBD and THC were taken out from the formulation. The cream will be applied twice daily.
  Interventions: Drug: OWC Control Cream

INTERVENTIONS:
Drug: OWC MGC cream — Topical cream containing 3% CBD and 3% THC for Psoriasis treatment
  Other Names: OWC psoriasis cream
  Arms: OWC MGC cream
Drug: OWC Control Cream — Topical Cream without active ingredients
  Arms: OWC Control Cream

SUMMARY:
This single center, prospective, double-blind, placebo-controlled, randomized two parts study (part I and part II) will assess the safety of topical cream (3% CBD and 3% THC), applied twice daily (bid), in healthy subjects, for up to 6 treatment weeks and additional 2 follow-up weeks.

DETAILED DESCRIPTION:
The study is divided into 2 stages. Healthy subjects will be consented to participate in the study.

Part I is designed to evaluate the single dose safety assessment of single application of MGC cream in 26 healthy volunteers (intact skin) for up to 24 consecutive hours under admission conditions in the clinical site. In this stage, the subjects will be divided into 3 application doses.

The following procedures will be performed:

* Time point 0- IV line, BP, Heart Rate, Blood testing (chemistry, blood count, Cannabinoids) and clinician evaluation of cannabis related psychological aspect (such as evaluation the cannabis abuse screening test).
* Time point 6 Hours- BP, Heart Rate Blood testing (chemistry, blood count, Cannabinoids)
* Time point 12- BP, Heart Rate, Blood testing (chemistry, blood count, Cannabinoids)
* Time point 24- BP, Heart Rate, Blood testing (chemistry, blood count, Cannabinoids) and and clinician evaluation of cannabis related psychological aspect (such as evaluation the cannabis abuse screening test).

Part II that will be followed the 24 hours (of part I) is designed to evaluate the repeated applications safety of MGC cream in healthy volunteers for up to 6 weeks, both in the clinic and by subjects at home.

20 healthy subjects that will be treated twice daily with:

* Maximal dose of 30 mg CBD : 30 mg THC, 1:1 ratio
* Placebo Control - 0 mg CBD : 0 mg THC, 1:1 ratio (vehicle)

This stage will be initiated at least 96 hour after completion part I of the study (washout period) .The placebo will be applied on one arm and the control on the second arm. Both, subject and investigator will be blinded as to the product/placebo allocation.

Application at home will be performed twice a day. Subjects will be asked to attend the clinic on day 0 of the part II treatment, once a week during the 6 weeks of daily application and 2 weeks post application. In each visit the following evaluations will be performed: BP, Heart Rate, Blood testing (chemistry, blood count, Cannabinoids) and clinician of cannabis related psychological aspect (such as evaluation the cannabis abuse screening test).

ELIGIBILITY:
Inclusion Criteria:

* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and electrocardiogram (ECGs).
* A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the OWC Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subjects with hemoglobin (Hb) values higher than ULN the normal range should always be excluded from enrollment.
* A female subject is eligible to participate if she is of non-childbearing potential (postmenopausal or pre-menopausal females with a documented tubal ligation or hysterectomy). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol.
* Agree not to participate in any other interventional clinical trials during the study
* Agree to follow study instructions meticulously

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Have evidence of significant, uncontrolled hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, gastrointestinal, or neurological disease. (Participants with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded).
* History of malignancy within 5 years of Screening or those with a strong family history of cancer (e.g., familial cancer disorders), with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated.
* A history of drug or alcohol abuse, or a history of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 mililiter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Consumption of: Barbiturates, Cocaine, Ethanol, SSRI's, Protease inhibitors, Warfarin, Sildenafil, Theophilline, Tricyclic antidepressants
* A positive test for human immunodeficiency virus (HIV) antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives (whichever is longer).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and OWC Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or OWC Medical Monitor, contraindicates their participation.
* Pregnant females as determined by positive urine human chorionic gonadotropin test at screening or prior to dosing.
* Are pregnant or nursing, or of child bearing potential and not practicing an effective means of birth control.
* Are not able to give adequate informed consent.
* Have any current problem or a history of substance abuse which, in the opinion of the investigator, might interfere with participation in the protocol.
* Have used marijuana within a month of starting the study.
* Fail the initial urine drug screen and blood test which tests for illicit drug use within the prior month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Incidence rate of AEs/ SAEs | 24 hours
  Collection of Adverse events and Serious Adverse Events
Incidence rate of AEs/ SAEs | 6 weeks
  Collection of Adverse events and Serious Adverse Events

SECONDARY OUTCOMES:
Specific AEs/ SAEs | Baseline to 24 hours
  Erythema Edema Swelling Itching Heat Pain Cellulitis Other
Specific AEs/ SAEs | baseline to 6 weeks
  Erythema Edema Swelling Itching Heat Pain Cellulitis Other

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No